CLINICAL TRIAL: NCT06457984
Title: Effects of Selenium Nutritional Supplement of Glucose, Nutritional Status, and Clinical Outcome Among Type 2 Diabetes Patients
Brief Title: Effects of Selenium Towards Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yu Kang, MD, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Selenium-T2DM-2024
Record Dates: First submitted 2024-05-08; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes
Keywords: selenium; intervention; glucose; nutritional status; clinical outcome
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Double(Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose selenium supplementation group+lifestyle intervention (Experimental): Low dose selenium supplementation:50μg/d +lifestyle intervention
  Interventions: Dietary Supplement: Selenium nutritional supplementation
- High dose selenium supplementation group+lifestyle intervention (Experimental): High dose selenium supplementation :300μg/d+lifestyle intervention
  Interventions: Dietary Supplement: Selenium nutritional supplementation
- Placebo control group+lifestyle intervention (Placebo Comparator): Placebo control group: sugar free chunk gum 1piles/d+lifestyle intervention
  Interventions: Dietary Supplement: Selenium nutritional supplementation

INTERVENTIONS:
Dietary Supplement: Selenium nutritional supplementation — Selenium yeast, as a safe from supplementation, could be a new nutritional intervention for lifecycle regulation of type 2 diabetes.
  Other Names: lifestyle intervention

SUMMARY:
According to the prevalence of non-communicable chronic diseases and aging population characteristics, this study is exploring the coexist effects combined with various dimensions: nutritional functions, metabolic homeostasis, inflammation and immunity by the selenium supplementation among type 2 diabetes, which based on insulin resistance, beta-cell function disorders, and body metabolic homeostasis disorders of the mechanism of type 2 diabetes by lifecycle so that could provide with a totally new and safe nutritional method for type 2 diabetes prevention and diagnosis.

DETAILED DESCRIPTION:
This study will last 16 weeks. There will be 300 subjects enrolled by random lottery methods in this randomized double-blind placebo-controlled clinical study by control group, low dose group and high dose group. During the study processing, follow-up visit by call, questionnaires, blood and stool collection, and functional testing will appear. Statistical analysis would be analysis according to the actual outcome of study.

ELIGIBILITY:
Inclusion Criteria:

.Range of age:18~75, both males and females are permitted.

.As to the diagnosis criteria of type 2 diabetes:glucose higher than 13.9mmol/L, drastic fluctuation (upper that 2mmol/L) , severe complication, or coupled with other severe chronic diseases( including overweight, obesity, lipid disorders, hypertension, ASCVD,HF, CKD, never appears.

.Treatments: exercise lifestyle intervention plus oral antidiabetic drugs, such as: single drug(metformin) plus exercise lifestyle intervention, coupled drugs(metformin+acarbose) plus exercise lifestyle intervention, both of them never use insulin.

.Signed with the informed consent, and enrolled in this study in volunteer.

Exclusion Criteria:

.Physical fitness must attach to the goal of Par-Q questionnaire and 6 minutes running test. Besides, individuals whose glucose has drastic fluctuation should be excluded.

.Coexist with severe complication and being in the urgent status during the progress of diseases, such as acute complication and infection, hyperplasia retinopathy, severe neuropathy, diabetic foot ulcer, coupled with cardiac insufficiency, diabetic massive proteinuria, recent myocardial infarction, cerebral infarction or cerebral hemorrhage, blood glucose higher than 13.9mmol/L or less than 3.9 mmol/L.

* Patients suffering various serious chronic diseases, including unstable angina, uncontrolled arrhythmia, severe valvular heart disease or cardiomyopathy;
* Uncontrolled hypertension or blood pressure over 180/110mmHg;

.In the period of trying to conceive or pregnant or lactating.

.Patients who have had cerebral infarction, stroke, history of major surgery, acute attack of infectious diseases or obvious sequelae of infection;

.Sever psychology disorders and mental diseases.

* The mass of selenium in body is over the upper limitation, or selenium yeast tablets, as a nutrition supplemented, subjects should not allergic to yeast, and cannot be included. Besides, patients who have recently taken selenium-rich health food or medicine;
* Severe malnutrition and overnutrition;
* Significant mobility and cognitive impairment;

.Sickle cell disease, hemodialysis, recent blood loss or blood transfusion, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The criteria about gender identity should be suit to the related legislation.
Enrollment: 300 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2025-05-07 (Estimated)

PRIMARY OUTCOMES:
Drugs of reduce glucose or stop using the antidiabetics. | 12 weeks
  Dose or types of antidiabetics drugs would reduce.

SECONDARY OUTCOMES:
GPX activity | 12 weeks
  Level of GPX-1 activity would decrease alone with the supplementation of selenium
Situation of glucose | 12 weeks
  Level of glucose would decrease alone with the supplementation of selenium
Nutrition status of selenium | 12 weeks
  Content of selenium in serum would increase alone with the supplementation of selenium
Status of immunity | 12 weeks
  Level of immunity indicator serum iron would increase along with the supplementation of selenium

CONTACTS AND LOCATIONS:
Overall Officials: yu kang, MD, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Yu Kang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Only be known by the research who do the work of random lottery method in this study.